CLINICAL TRIAL: NCT05160311
Title: Percutaneous Revascularization in Infarction With Late Presentation and Absence of Viability: Effects on Left Ventricular Remodeling and Contractility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Barbara Porto Valente, Cardiology Physician, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5106
Record Dates: First submitted 2021-10-29; First posted 2021-12-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Myocardial Dysfunction; Percutaneous Coronary Intervention
Keywords: STEMI; myocardial viability; Late percutaneous coronary intervention; myocardial remodelling; Myocardial reperfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Drug-Eluting Stents; Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: Patients who had underestimated STEMI with more than 24 hours up to 28 days referred by the Cross System (Central For Regulation of Health Services Supply) and the Campo Limpo Hospital (Co-participant Center) will be admitted sequentially for coronary angiography in the hemodynamics sector of the Instituto Dante Pazzanese de Cardiologia (IDPC) from August 2021 to February 2023.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized Medical Treatment (OMT) (Other): The patient considered non-viable by MRI and randomized to Optimized Medical Treatment (OMT) will be treated according to Optimized Medical Treatment guidelines for Coronary Artery Disease (CAD)
  Interventions: Drug: Optimized Medical Treatment (OMT)
- Angioplasty (PCI) and Optimized Medical Treatment (OMT) (Experimental): The patient considered non-viable and randomized to Coronary Angioplasty will be treated with drug-eluting stent (PCI) and Optimized Medical Treatment (OMT)
  Interventions: Drug: Optimized Medical Treatment (OMT); Device: Drug Eluting Stent (DES) Coronary Angioplasty

INTERVENTIONS:
Drug: Optimized Medical Treatment (OMT) — Optimized Medical Drug Treatment
Device: Drug Eluting Stent (DES) Coronary Angioplasty — Percutaneous Angioplasty with DES
  Arms: Angioplasty (PCI) and Optimized Medical Treatment (OMT)

SUMMARY:
The purpose of this study is to evaluate whether late recanalization in patients with ST elevation myocardial infarction (STEMI) without Viability on Cardiovascular Magnetic Resonance Image (MRI) can reduce the reverse remodeling through the reduction of the End Systolic Volume (ESV) at 6 months.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether late recanalization in patients with ST elevation myocardial infarction (STEMI) without Viability on Cardiovascular Magnetic Resonance can reduce the reverse remodeling through the reduction of the End Systolic Volume (ESV) at 6 months and through the improvement in segmental contractility of infarcted related artery at MRI.

ELIGIBILITY:
Inclusion Criteria

1. STEMI not reperfused between 24 hours and 28 days
2. MI-related artery with > or = 50%
3. Segmental dysfunction in the artery related to infarction.
4. Technical feasibility for PCI recanalization
5. Absence of Myocardial Viability

3.3 Exclusion criteria

1. Age > 80 years
2. < 1 year life expectancy
3. Post MI Angina
4. Clinical Instability
5. Electrical Instability
6. Previous Infarction with segment disfunction
7. New York Heart Association (NYHA) class III or IV of heart failure.
8. Previous diagnosis of congestive heart failure or cardiomyopathy
9. Severe heart valve disease
10. Absence of segmental dysfunction in the artery related to infarction
11. Coronary angiography without obstructive lesions
12. Indication of myocardial revascularization surgery
13. Opted for clinical treatment for technical reasons
14. Serum creatinine concentration greater than 2.5 mg/dl
15. Pacemaker or Implantable Cardiodefibrillator (ICD)
16. Brain Clip Carriers
17. Patients with Cochlear Implants
18. Refusal to sign the Informed Consent Form (ICF).
19. Inability to maintain outpatient follow-up for 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Reverse myocardial remodeling after late recanalization in patients without viability | 6 months
  Evaluate reverse remodeling after late recanalization in patients without viability measuring End Systolic Volume (ESV) by MRI

SECONDARY OUTCOMES:
Assessement of Left Ventricle Ejection Fraction (LVEF) | 6 months
  Change in LVEF measured by MRI The degree of LVEF recovery after a MI provides important prognostic information. Patients with no recovery in LVEF after MI are at high risk of sudden cardiac arrest events and death.
Assessement of Myocardial contractility | 6 months
  Evaluate the change of reverse LV remodeling after late recanalization assessed by MRI.
Evaluate Quality of Life | 6 months
  Evaluate change from baseline in patients Quality of life using Abbreviated World Health Organization Quality of Life (WHOQOL-BREF) questionnaire.
  The WHOQOL-Bref (Field Trial Version) produces a profile with four domain scores and two individually scored items about an individual's overall perception of quality of life and health. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. The possible raw score ranges for each domain are as follows: Physical Health=28, Psychological=24, Social Relationships=12, and Environment=32.
Acute MI Event | 6 months
  Incidence of Acute Myocardial Infarct.
Unplanned revascularization (Ischemia Driven and Not Ischemia Driven) | 6 months
  Incidence of Unplanned Myocardial revascularization (Ischemia Driven and Not Ischemia Driven) after hospital discharge
Cardiovascular Death | 6 months
  Incidence of Cardiovascular Death. Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality, cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
Cardiovascular-Related Hospitalization | 6 months
  Incidence of New Cardiovascular related Hospitalization after discharge
Stroke Event | 6 months
  Incidence of Stroke Event Stroke is defined as the rapid onset of a new persistent neurologic deficit attributed to an obstruction in cerebral blood flow and/or cerebral hemorrhage with no apparent non-vascular cause (e.g., trauma, tumor, or infection).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Valente, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long-term effects of intravenous thrombolysis in acute myocardial infarction: final report of the GISSI study. Gruppo Italiano per lo Studio della Streptochi-nasi nell'Infarto Miocardico (GISSI). Lancet. 1987 Oct 17;2(8564):871-4. PMID 2889079
- [Background] O'Neill W, Timmis GC, Bourdillon PD, Lai P, Ganghadarhan V, Walton J Jr, Ramos R, Laufer N, Gordon S, Schork MA, et al. A prospective randomized clinical trial of intracoronary streptokinase versus coronary angioplasty for acute myocardial infarction. N Engl J Med. 1986 Mar 27;314(13):812-8. doi: 10.1056/NEJM198603273141303. PMID 2936956
- [Background] Piegas LS, Feitosa G, Mattos LA, Nicolau JC, Rossi Neto JM et al. Brazilian Society of Cardiology. IV Guideline of the Brazilian Society of Cardiology on The Treatment of Acute Myocardial Infarction with ST Segment Supradeslevel. Arq Bras Cardiol.2009;93(6 supl.2):e179-e264.
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Eagle KA, Goodman SG, Avezum A, Budaj A, Sullivan CM, Lopez-Sendon J; GRACE Investigators. Practice variation and missed opportunities for reperfusion in ST-segment-elevation myocardial infarction: findings from the Global Registry of Acute Coronary Events (GRACE). Lancet. 2002 Feb 2;359(9304):373-7. doi: 10.1016/S0140-6736(02)07595-5. PMID 11844506
- [Background] Cohen M, Gensini GF, Maritz F, Gurfinkel EP, Huber K, Timerman A, Krzeminska-Pakula M, Santopinto J, Hecquet C, Vittori L; TETAMI Investigators. Prospective evaluation of clinical outcomes after acute ST-elevation myocardial infarction in patients who are ineligible for reperfusion therapy: preliminary results from the TETAMI registry and randomized trial. Circulation. 2003 Oct 21;108(16 Suppl 1):III14-21. doi: 10.1161/01.CIR.0000091832.74006.1C. PMID 14605015
- [Background] Late Assessment of Thrombolytic Efficacy (LATE) study with alteplase 6-24 hours after onset of acute myocardial infarction. Lancet. 1993 Sep 25;342(8874):759-66. PMID 8103874
- [Background] Dzavik V, Beanlands DS, Davies RF, Leddy D, Marquis JF, Teo KK, Ruddy TD, Burton JR, Humen DP. Effects of late percutaneous transluminal coronary angioplasty of an occluded infarct-related coronary artery on left ventricular function in patients with a recent (< 6 weeks) Q-wave acute myocardial infarction (Total Occlusion Post-Myocardial Infarction Intervention Study [TOMIIS]--a pilot study). Am J Cardiol. 1994 May 1;73(12):856-61. doi: 10.1016/0002-9149(94)90809-5. PMID 8184807
- [Background] Yousef ZR, Marber MS. The open artery hypothesis: potential mechanisms of action. Prog Cardiovasc Dis. 2000 May-Jun;42(6):419-38. PMID 10871164
- [Background] Horie H, Takahashi M, Minai K, Izumi M, Takaoka A, Nozawa M, Yokohama H, Fujita T, Sakamoto T, Kito O, Okamura H, Kinoshita M. Long-term beneficial effect of late reperfusion for acute anterior myocardial infarction with percutaneous transluminal coronary angioplasty. Circulation. 1998 Dec 1;98(22):2377-82. doi: 10.1161/01.cir.98.22.2377. PMID 9832481
- [Background] Yousef ZR, Redwood SR, Bucknall CA, Sulke AN, Marber MS. Late intervention after anterior myocardial infarction: effects on left ventricular size, function, quality of life, and exercise tolerance: results of the Open Artery Trial (TOAT Study). J Am Coll Cardiol. 2002 Sep 4;40(5):869-76. doi: 10.1016/s0735-1097(02)02058-2. PMID 12225709
- [Background] Silva JC, Rochitte CE, Junior JS, Tsutsui J, Andrade J, Martinez EE, Moffa PJ, Menegheti JC, Kalil-Filho R, Ramires JF, Nicolau JC. Late coronary artery recanalization effects on left ventricular remodelling and contractility by magnetic resonance imaging. Eur Heart J. 2005 Jan;26(1):36-43. doi: 10.1093/eurheartj/ehi011. Epub 2004 Nov 29. PMID 15615797
- [Background] Hochman JS, Lamas GA, Buller CE, Dzavik V, Reynolds HR, Abramsky SJ, Forman S, Ruzyllo W, Maggioni AP, White H, Sadowski Z, Carvalho AC, Rankin JM, Renkin JP, Steg PG, Mascette AM, Sopko G, Pfisterer ME, Leor J, Fridrich V, Mark DB, Knatterud GL; Occluded Artery Trial Investigators. Coronary intervention for persistent occlusion after myocardial infarction. N Engl J Med. 2006 Dec 7;355(23):2395-407. doi: 10.1056/NEJMoa066139. Epub 2006 Nov 14. PMID 17105759
- [Background] Abbate A, Biondi-Zoccai GG, Appleton DL, Erne P, Schoenenberger AW, Lipinski MJ, Agostoni P, Sheiban I, Vetrovec GW. Survival and cardiac remodeling benefits in patients undergoing late percutaneous coronary intervention of the infarct-related artery: evidence from a meta-analysis of randomized controlled trials. J Am Coll Cardiol. 2008 Mar 4;51(9):956-64. doi: 10.1016/j.jacc.2007.11.062. Epub 2008 Feb 6. PMID 18308165
- [Background] Sabate M. Revascularization of the infarct-related artery: never too late to do well. J Am Coll Cardiol. 2008 Mar 4;51(9):965-7. doi: 10.1016/j.jacc.2008.01.003. Epub 2008 Feb 5. No abstract available. PMID 18308166
- [Background] Erne P, Schoenenberger AW, Burckhardt D, Zuber M, Kiowski W, Buser PT, Dubach P, Resink TJ, Pfisterer M. Effects of percutaneous coronary interventions in silent ischemia after myocardial infarction: the SWISSI II randomized controlled trial. JAMA. 2007 May 9;297(18):1985-91. doi: 10.1001/jama.297.18.1985. PMID 17488963
- [Background] Allman KC, Shaw LJ, Hachamovitch R, Udelson JE. Myocardial viability testing and impact of revascularization on prognosis in patients with coronary artery disease and left ventricular dysfunction: a meta-analysis. J Am Coll Cardiol. 2002 Apr 3;39(7):1151-8. doi: 10.1016/s0735-1097(02)01726-6. PMID 11923039
- [Background] Udelson JE, Pearte CA, Kimmelstiel CD, Kruk M, Kufera JA, Forman SA, Teresinska A, Bychowiec B, Marin-Neto JA, Hochtl T, Cohen EA, Caramori P, Busz-Papiez B, Adlbrecht C, Sadowski ZP, Ruzyllo W, Kinan DJ, Lamas GA, Hochman JS. The Occluded Artery Trial (OAT) Viability Ancillary Study (OAT-NUC): influence of infarct zone viability on left ventricular remodeling after percutaneous coronary intervention versus optimal medical therapy alone. Am Heart J. 2011 Mar;161(3):611-21. doi: 10.1016/j.ahj.2010.11.020. PMID 21392619
- [Background] Bellenger NG, Yousef Z, Rajappan K, Marber MS, Pennell DJ. Infarct zone viability influences ventricular remodelling after late recanalisation of an occluded infarct related artery. Heart. 2005 Apr;91(4):478-83. doi: 10.1136/hrt.2004.034918. PMID 15772205
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] Selvanayagam JB, Kardos A, Francis JM, Wiesmann F, Petersen SE, Taggart DP, Neubauer S. Value of delayed-enhancement cardiovascular magnetic resonance imaging in predicting myocardial viability after surgical revascularization. Circulation. 2004 Sep 21;110(12):1535-41. doi: 10.1161/01.CIR.0000142045.22628.74. Epub 2004 Sep 7. PMID 15353496
- [Background] Camici PG, Prasad SK, Rimoldi OE. Stunning, hibernation, and assessment of myocardial viability. Circulation. 2008 Jan 1;117(1):103-14. doi: 10.1161/CIRCULATIONAHA.107.702993. No abstract available. PMID 18172050
- [Background] Romero J, Xue X, Gonzalez W, Garcia MJ. CMR imaging assessing viability in patients with chronic ventricular dysfunction due to coronary artery disease: a meta-analysis of prospective trials. JACC Cardiovasc Imaging. 2012 May;5(5):494-508. doi: 10.1016/j.jcmg.2012.02.009. PMID 22595157
- [Background] Gerber BL, Rousseau MF, Ahn SA, le Polain de Waroux JB, Pouleur AC, Phlips T, Vancraeynest D, Pasquet A, Vanoverschelde JL. Prognostic value of myocardial viability by delayed-enhanced magnetic resonance in patients with coronary artery disease and low ejection fraction: impact of revascularization therapy. J Am Coll Cardiol. 2012 Feb 28;59(9):825-35. doi: 10.1016/j.jacc.2011.09.073. PMID 22361403
- [Background] STATACorp. 2019. Stata Statistical Software: Release 16.0. College Station, Texas : Stata Corporation